CLINICAL TRIAL: NCT05892549
Title: COVID-19: Early Detection of Worsening by Voice and Respiratory Pattern Characteristics
Acronym: COVOICE
Status: Recruiting | Type: Observational
Sponsor: Direction Centrale du Service de Santé des Armées (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-COVID19-21; 2020-A03182-37 (Other: IDRCB)
Record Dates: First submitted 2023-06-06; First posted 2023-06-07 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Sars-CoV-2 Infection; COVID-19
Keywords: Voice
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- COVID
  Interventions: Device: COVOICE application use - follow-up
- Other respiratory diseases
  Interventions: Device: COVOICE application use - follow-up
- Healthy
  Interventions: Device: COVOICE application use - initial

INTERVENTIONS:
Device: COVOICE application use - initial — Recording (only once) of sound related to respiratory movements, coughing and voice using a mobile phone application
  Groups: Healthy
Device: COVOICE application use - follow-up — Daily recording of sound related to respiratory movements, coughing and voice using a mobile phone application. Duration: up to 30 days
  Groups: COVID; Other respiratory diseases

SUMMARY:
In some clinical forms of COVID-19, an uncontrolled hyper-inflammatory reaction known as a "cytokine storm" appears abruptly, around day 7, and is associated with rapid respiratory deterioration, requiring hospitalization in an intensive care unit (ICU).

At present, although risk factors for this severe form have been described, there are no validated criteria for determining which individual patients will develop this aggravation.

The study of respiratory sounds (amplitude, frequency, ...) has made it possible in other respiratory pathologies (e.g., chronic obstructive pulmonary disease) to predict exacerbations several days in advance.

Having a predictive respiratory pattern for worsening in COVID-19 would make it possible to anticipate the need for intensive care hospital beds, by means of a tool easily available on a mobile phone.

ELIGIBILITY:
Inclusion Criteria:

* French speaking
* Affiliated to a social security system
* Owning a mobile phone capable of accessing the COVOICE application

Exclusion Criteria:

* Incapable adults
* People deprived of their liberty
* People under administrative or judicial supervision
* Patients intubated or hospitalized in intensive care unit

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study population is composed of people coming to a hospital or to a COVID screening center.
Sampling Method: Non-Probability Sample
Enrollment: 1188 (Estimated)
Dates: Start 2023-06-12 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Sensitivity of the respiratory pattern demonstrated in the COVID patients who experienced respiratory worsening | Through study completion (36 months)
Specificity of the respiratory pattern demonstrated in the COVID patients who experienced respiratory worsening | Through study completion (36 months)

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital d'Instruction des Armées Bégin, Saint-Mandé, France

IPD SHARING:
Plan to Share IPD: Undecided